CLINICAL TRIAL: NCT00152529
Title: "C.A.T.C.H.-I.T." Competent Adulthood Transition With Cognitive, Humanistic and Interpersonal Teaching
Brief Title: C.A.T.C.H.-I.T.Competent Adulthood Transition With Cognitive, Humanistic and Interpersonal Teaching
Status: Terminated | Type: Observational
Why Stopped: Study completed
Sponsor: University of Chicago (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 12591A; U48/CCU309674 - 12591A
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Depression
Keywords: Depression, educational site for depression
MeSH Terms: conditions — Depression | interventions — Mass Screening

INTERVENTIONS:
Behavioral: Screening (Behavior)

SUMMARY:
The purpose of this study is to adapt depression prevention interventions of proven benefit to the primary care setting in a manner that would be acceptable and potentially available to young adults in the community.

DETAILED DESCRIPTION:
Our study goal is to develop a prototype combination primary care-web based depression intervention for young adults ages 18-24years in urban community and university settings. The content development will include: (1) two brief (15 minutes) primary care counseling sessions, (2) one introductory web based module, (3) four web-based cognitive behavior teaching modules, (4) three web-based modules discussing relationship building skills (IPT), and (5) a final web module discussing self-recognition, evidence-based treatment, and stigma. Eight young adult volunteers will evaluate the program in three loops of evaluation and revision in a modified focus group approach. This protocol was approved by the Johns Hopkins Joint Committee on Clinical Investigations.

Primary Outcomes:

The primary outcome variables relate to the functionality and acceptability of the intervention. These variables include readability, ease of understanding, acceptability, and helpfulness of each component of the intervention, and a global rating of each

Secondary Outcomes:

Process measures (time on site, exercise completion), outcomes (mood and intermediate outcomes-social adjustment, dysfunctional thinking), and knowledge and opinions of current treatments for depression. These data will be helpful in planning for a future Focus groups of 5-10 individuals have been used successfully to provide initial product evaluations or to develop general themes in attitude research. Summary statistics will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria include being between ages 18-24 and having a family history of depression. Preference will be given in selection of participants to those of who have not been treated for depression in the past.

Exclusion Criteria:

* Moderate or greater risk of having depression (CESD score > 16) or current treatment for depression. Those who have a history of past treatment of depression will not be excluded.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8
Dates: Start 2003-10; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin W Van Voorhees, MD, Principal Investigator — The University of Chicago, 5841 South Maryland Ave., MC 2007 Chicago, IL 60637
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Eisen JC, Marko-Holguin M, Fogel J, Cardenas A, Bahn M, Bradford N, Fagan B, Wiedmann P, Van Voorhees BW. Pilot Study of Implementation of an Internet-Based Depression Prevention Intervention (CATCH-IT) for Adolescents in 12 US Primary Care Practices: Clinical and Management/Organizational Behavioral Perspectives. Prim Care Companion CNS Disord. 2013;15(6):PCC.10m01065. doi: 10.4088/PCC.10m01065. Epub 2013 Dec 19. PMID 24800110
- [Derived] Hoek W, Marko M, Fogel J, Schuurmans J, Gladstone T, Bradford N, Domanico R, Fagan B, Bell C, Reinecke MA, Van Voorhees BW. Randomized controlled trial of primary care physician motivational interviewing versus brief advice to engage adolescents with an Internet-based depression prevention intervention: 6-month outcomes and predictors of improvement. Transl Res. 2011 Dec;158(6):315-25. doi: 10.1016/j.trsl.2011.07.006. Epub 2011 Aug 19. PMID 22061038
- [Derived] Iloabachie C, Wells C, Goodwin B, Baldwin M, Vanderplough-Booth K, Gladstone T, Murray M, Fogel J, Van Voorhees BW. Adolescent and parent experiences with a primary care/Internet-based depression prevention intervention (CATCH-IT). Gen Hosp Psychiatry. 2011 Nov-Dec;33(6):543-55. doi: 10.1016/j.genhosppsych.2011.08.004. Epub 2011 Sep 28. PMID 21958447